CLINICAL TRIAL: NCT04332614
Title: Email Campaign to Encourage Patients to Complete Sign-up Process for Geisinger's Patient Portal
Brief Title: Email Campaign to Increase Uptake of myGeisinger
Status: Completed | Type: Observational
Sponsor: Geisinger Clinic (Other)
Responsible Party: Principal Investigator, Amir Goren, Program Director, Behavioral Insights Team, Geisinger Clinic
Other Study IDs: 2020-0315
Record Dates: First submitted 2020-03-31; First posted 2020-04-02 (Actual); Results first posted 2021-05-03 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Telehealth; Health Behavior
Keywords: Behavioral Economics; Patient Portal; Social Proof; Endowment Effect; Less-is-better
MeSH Terms: conditions — Health Behavior | interventions — Financial Management

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Control: A standard marketing message encouraging activation and describing the benefits of myGeisinger
  Interventions: Behavioral: Standard email
- Focused on provider communication: A simple message focused on one benefit of myGeisinger: communicating easily with providers
  Interventions: Behavioral: Less-is-better
- Focused on scheduling: A simple message focused on one benefit of myGeisinger: scheduling and managing appointments online
  Interventions: Behavioral: Less-is-better
- Focused on medical information access: A simple message focused on one benefit of myGeisinger: accessing medical information, like test results
  Interventions: Behavioral: Less-is-better
- Social proof: A message similar to control, but including information about how many other patients are using myGeisinger
  Interventions: Behavioral: Social proof
- Endowment / decision staging: A message similar to control, but framing myGeisinger as something that patients already have, and just need to take one more step to activate.
  Endowment: Give patients the impression they already have the account, so they value it more.
  Decision staging: Break down the process into multiple stages - "having" an account and "activating" that account- and giving the impression that they are almost there because the first stage is complete
  Interventions: Behavioral: Endowment / decision staging

INTERVENTIONS:
Behavioral: Less-is-better — Email
  Groups: Focused on medical information access; Focused on provider communication; Focused on scheduling
Behavioral: Social proof — Email
  Groups: Social proof
Behavioral: Endowment / decision staging — Email
  Groups: Endowment / decision staging
Behavioral: Standard email — Email
  Groups: Control

SUMMARY:
The purpose of the current study is to test different email messages to determine the most effect way of promoting enrollment in Geisinger's patient portal, called myGeisinger.

DETAILED DESCRIPTION:
Online patient portals are convenient tools that improve patient access to healthcare services while often reducing burden to both patients and providers. However, fewer than half of patients have enrolled in Geisinger's patient portal, myGeisinger.

The purpose of the current study is to assess what kind of messaging improves the effectiveness of an email campaign targeted at enrolling patients into Geisinger's online patient portal, called myGeisinger. Currently, Geisinger sends an email every month to patients who have started but not completed the enrollment process (they have had an activation code generated but have not yet used that code to enroll). This study will A/B test 5 email messages to assess if they perform better than the current standard email message.

Performance will be assessed based on whether patients open the email, click on the myGeisinger enrollment link, and enroll in myGeisinger. Statistical analyses will employ generalized linear models with a binary distribution and log-link function.

ELIGIBILITY:
Inclusion Criteria:

* Geisinger patients whose myGeisinger status is "Pending", meaning an activation code has been generated for them, but they have not completed activation

Exclusion Criteria:

* Patients without email addresses on file
* Patients who received emails from this monthly myGeisinger marketing campaign within the last 2 months

Ages: 18 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population consists of Geisinger patients whose myGeisinger status is "Pending" and who have an email address on file.
Sampling Method: Probability Sample
Enrollment: 14099 (Actual)
Dates: Start 2020-04-06 (Actual); Primary Completion 2020-04-13 (Actual); Study Completion 2020-05-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amir Goren, PhD, Principal Investigator — Geisinger Clinic
Locations (1):
- Geisinger, Danville, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Data with no personally identifiable information will be made available to other researchers on the Open Science Framework for transparency. This will include the essential data and code needed to replicate the analysis that yielded reported findings.
Supporting Information: Analytic Code
Time Frame: The data will become available after publication of study results in a scientific journal and will be available as long as the Open Science Framework hosts the data.
Access Criteria: The data on the Open Science Framework will be open to anyone requesting that information.
URL: http://osf.io

RESULTS

PARTICIPANT FLOW:
Groups:
- Endowment / Decision Staging: A message similar to control, but framing myGeisinger as something that patients already have, and just need to take one more step to activate.
  Endowment: Give patients the impression they already have the account, so they value it more.
  Decision staging: Break down the process into multiple stages - "having" an account and "activating" that account- and giving the impression that they are almost there because the first stage is complete
  Endowment / decision staging: Email
Period: ~1 Week After Study Launch
Arm/Group | Control | Focused on Provider Communication | Focused on Scheduling | Focused on Medical Information Access | Social Proof | Endowment / Decision Staging
Started (Randomized and attempted to email) | 2350 | 2350 | 2350 | 2350 | 2350 | 2349
Data in EHR (Patient was found in Electronic Health Record ~1 week after intervention) | 2245 | 2273 | 2251 | 2254 | 2251 | 2249
Completed (Email delivered (did not bounce back)) | 2117 | 2129 | 2124 | 2131 | 2127 | 2115
Not Completed | 233 | 221 | 226 | 219 | 223 | 234
Period: ~1 Month After Study Launch
Arm/Group | Control | Focused on Provider Communication | Focused on Scheduling | Focused on Medical Information Access | Social Proof | Endowment / Decision Staging
Started | 2117 | 2129 | 2124 | 2131 | 2127 | 2115
Completed (Record was found in EHR ~1 month after intervention AND email was delivered (did not bounce back)) | 2095 | 2107 | 2094 | 2107 | 2107 | 2096
Not Completed | 22 | 22 | 30 | 24 | 20 | 19

BASELINE CHARACTERISTICS:
Population: Investigators did not have access to baseline demographic information for study participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Focused on Provider Communication | Focused on Scheduling | Focused on Medical Information Access | Social Proof | Endowment / Decision Staging | Total
Number analyzed (Participants) | 2350 | 2350 | 2350 | 2350 | 2350 | 2349 | 14099
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | NA — Data not collected | NA — Data not collected | NA — Data not collected | NA — Data not collected | NA — Data not collected | NA — Data not collected | NA — Total not calculated because data are not available (NA) in one or more arms.
  Between 18 and 65 years | NA — Data not collected | NA — Data not collected | NA — Data not collected | NA — Data not collected | NA — Data not collected | NA — Data not collected | NA — Total not calculated because data are not available (NA) in one or more arms.
  >=65 years | NA — Data not collected | NA — Data not collected | NA — Data not collected | NA — Data not collected | NA — Data not collected | NA — Data not collected | NA — Total not calculated because data are not available (NA) in one or more arms.
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | NA — Data not collected | NA — Data not collected | NA — Data not collected | NA — Data not collected | NA — Data not collected | NA — Data not collected | NA — Total not calculated because data are not available (NA) in one or more arms.
  Male | NA — Data not collected | NA — Data not collected | NA — Data not collected | NA — Data not collected | NA — Data not collected | NA — Data not collected | NA — Total not calculated because data are not available (NA) in one or more arms.
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 2350 | 2350 | 2350 | 2350 | 2350 | 2349 | 14099

OUTCOME MEASURES:

1. Primary Outcome: Email Opened: Control vs. Less-is-better vs. Social Proof vs. Endowment
Description: Whether email was opened (yes / no)
Time Frame: 8-10 days post-intervention
Population: Patients who were delivered an email (i.e. email did not bounce back) and for whom there was a record in the EHR 10 days post-intervention.
Measure: Count of Participants; unit: Participants
Groups:
- Less-is-better: A simple message focused on one benefit of myGeisinger.
Arm/Group | Control | Less-is-better | Social Proof | Endowment / Decision Staging
Number analyzed (Participants) | 2117 | 6384 | 2127 | 2115
Participants | 558 | 1528 | 375 | 488
Statistical Analysis 1: Comparison: Control vs Less-is-better; Test type: Superiority; p = 0.0248, Regression, Logistic — We used an a priori threshold of p < .05. All 3 comparisons run within same logistic regression model; Odds Ratio (OR) = 0.8791371, 95% CI 2-sided [0.7856042 to 0.9838058]
Statistical Analysis 2: Comparison: Control vs Social Proof; Test type: Superiority; p < 0.0001, Regression, Logistic — We used an a priori threshold of p < .05. All 3 comparisons run within same logistic regression model; Odds Ratio (OR) = 0.5980109, 95% CI 2-sided [0.5159511 to 0.6931219]
Statistical Analysis 3: Comparison: Control vs Endowment / Decision Staging; Test type: Superiority; p = 0.0133, Regression, Logistic — We used an a priori threshold of p < .05. All 3 comparisons run within same logistic regression model; Odds Ratio (OR) = 0.8380003, 95% CI 2-sided [0.7285712 to 0.9638653]

2. Primary Outcome: Link Clicked: Control vs. Less-is-better vs. Social Proof vs. Endowment
Description: Whether the link / button to start the activation process was clicked (yes / no)
Time Frame: 8-10 days post-intervention
Population: Patients who opened the intervention email and for whom there was a record in the EHR 10 days post-intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Less-is-better | Social Proof | Endowment / Decision Staging
Number analyzed (Participants) | 558 | 1528 | 375 | 488
Participants | 134 | 160 | 31 | 73
Statistical Analysis 1: Comparison: Control vs Less-is-better; Test type: Superiority; p < 0.0001, Regression, Logistic — We used an a priori threshold of p < .05. All 3 comparisons run within same logistic regression model; Odds Ratio (OR) = 0.3700794, 95% CI 2-sided [0.2870513 to 0.4771231]
Statistical Analysis 2: Comparison: Control vs Social Proof; Test type: Superiority; p < 0.0001, Regression, Logistic — We used an a priori threshold of p < .05. All 3 comparisons run within same logistic regression model; Odds Ratio (OR) = 0.2851440, 95% CI 2-sided [0.1881589 to 0.4321194]
Statistical Analysis 3: Comparison: Control vs Endowment / Decision Staging; Test type: Superiority; p = 0.0003, Regression, Logistic — We used an a priori threshold of p < .05. All 3 comparisons run within same logistic regression model; Odds Ratio (OR) = 0.5565905, 95% CI 2-sided [0.4059477 to 0.7631354]

3. Primary Outcome: Enrollment: Control vs. Less-is-better vs. Social Proof vs. Endowment
Description: Whether the patient enrolled in myGeisinger (yes / no)
Time Frame: 8-10 days post-intervention
Population: Patients who opened the intervention email and for whom there was a record in the EHR 10 days post-intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Less-is-better | Social Proof | Endowment / Decision Staging
Number analyzed (Participants) | 558 | 1528 | 375 | 488
Participants | 41 | 83 | 18 | 38
Statistical Analysis 1: Comparison: Control vs Less-is-better; Test type: Superiority; p = 0.103, Regression, Logistic — We used an a priori threshold of p < .05. All 3 comparisons run within same logistic regression model; Odds Ratio (OR) = 0.72429741, 95% CI 2-sided [0.49167734 to 1.0669736]
Statistical Analysis 2: Comparison: Control vs Social Proof; Test type: Superiority; p = 0.120, Regression, Logistic — We used an a priori threshold of p < .05. All 3 comparisons run within same logistic regression model; Odds Ratio (OR) = 0.63578603, 95% CI 2-sided [0.35943749 to 1.1246013]
Statistical Analysis 3: Comparison: Control vs Endowment / Decision Staging; Test type: Superiority; p = 0.789, Regression, Logistic — We used an a priori threshold of p < .05. All 3 comparisons run within same logistic regression model; Odds Ratio (OR) = 1.06482385, 95% CI 2-sided [0.67282661 to 1.6852036]

4. Secondary Outcome: Email Opened: Control vs. Less-is-better vs. Social Proof vs. Endowment
Description: Whether email was opened (yes / no)
Time Frame: 32-35 days post-intervention
Population: Patients who were delivered an email (i.e. email did not bounce back) and for whom there was a record in the EHR 32 days post-intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Less-is-better | Social Proof | Endowment / Decision Staging
Number analyzed (Participants) | 2095 | 6308 | 2107 | 2096
Participants | 591 | 1626 | 402 | 512
Statistical Analysis 1: Comparison: Control vs Less-is-better; Test type: Superiority; p = 0.0286, Regression, Logistic — We used an a priori threshold of p < .05. All 3 comparisons run within same logistic regression model; Odds Ratio (OR) = 0.8837908, 95% CI 2-sided [0.7912382 to 0.9871694]
Statistical Analysis 2: Comparison: Control vs Social Proof; Test type: Superiority; p < 0.0001, Regression, Logistic — We used an a priori threshold of p < .05. All 3 comparisons run within same logistic regression model; Odds Ratio (OR) = 0.6000149, 95% CI 2-sided [0.5193168 to 0.6932528]
Statistical Analysis 3: Comparison: Control vs Endowment / Decision Staging; Test type: Superiority; p = 0.0055, Regression, Logistic; Odds Ratio (OR) = 0.8225743, 95% CI 2-sided [0.7167043 to 0.9440832]

5. Secondary Outcome: Link Clicked: Control vs. Less-is-better vs. Social Proof vs. Endowment
Description: Whether the link / button to start the activation process was clicked (yes / no)
Time Frame: 32-35 days post-intervention
Population: Patients who opened the intervention email and for whom there was a record in the EHR 32 days post-intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Less-is-better | Social Proof | Endowment / Decision Staging
Number analyzed (Participants) | 591 | 1626 | 402 | 512
Participants | 147 | 188 | 34 | 86
Statistical Analysis 1: Comparison: Control vs Less-is-better; Test type: Superiority; p < 0.0001, Regression, Logistic — We used an a priori threshold of p < .05. All 3 comparisons run within same logistic regression model; Odds Ratio (OR) = 0.3948795, 95% CI 2-sided [0.3104370 to 0.5022914]
Statistical Analysis 2: Comparison: Control vs Social Proof; Test type: Superiority; p < 0.0001, Regression, Logistic — We used an a priori threshold of p < .05. All 3 comparisons run within same logistic regression model; Odds Ratio (OR) = 0.2790595, 95% CI 2-sided [0.1875017 to 0.4153254]
Statistical Analysis 3: Comparison: Control vs Endowment / Decision Staging; Test type: Superiority; p = 0.0011, Regression, Logistic — We used an a priori threshold of p < .05. All 3 comparisons run within same logistic regression model; Odds Ratio (OR) = 0.6097538, 95% CI 2-sided [0.4528751 to 0.8209762]

6. Secondary Outcome: Enrollment: Control vs. Less-is-better vs. Social Proof vs. Endowment
Description: Whether the patient enrolled in myGeisinger (yes / no)
Time Frame: 32-35 days post-intervention
Population: Patients who opened the intervention email and for whom there was a record in the EHR 32 days post-intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Less-is-better | Social Proof | Endowment / Decision Staging
Number analyzed (Participants) | 591 | 1626 | 402 | 512
Participants | 55 | 152 | 29 | 55
Statistical Analysis 1: Comparison: Control vs Less-is-better; Test type: Superiority; p = 0.976, Regression, Logistic — We used an a priori threshold of p < .05. All 3 comparisons run within same logistic regression model; Odds Ratio (OR) = 1.0049587, 95% CI 2-sided [0.72693253 to 1.3893201]
Statistical Analysis 2: Comparison: Control vs Social Proof; Test type: Superiority; p = 0.246, Regression, Logistic — We used an a priori threshold of p < .05. All 3 comparisons run within same logistic regression model; Odds Ratio (OR) = 0.7576895, 95% CI 2-sided [0.47412590 to 1.2108458]
Statistical Analysis 3: Comparison: Control vs Endowment / Decision Staging; Test type: Superiority; p = 0.428, Regression, Logistic — We used an a priori threshold of p < .05. All 3 comparisons run within same logistic regression model; Odds Ratio (OR) = 1.1728665, 95% CI 2-sided [0.79090107 to 1.7393021]

7. Secondary Outcome: Email Opened: Within Less-is-better (Provider Communication vs. Managing Appointments vs. Medical Information Access)
Description: Whether email was opened (yes / no)
Time Frame: 8-10 days post-intervention
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Focused on Provider Communication | Focused on Scheduling | Focused on Medical Information Access
Number analyzed (Participants) | 2129 | 2124 | 2131
Participants | 524 | 522 | 482
Statistical Analysis 1: Comparison: Focused on Provider Communication vs Focused on Scheduling; Test type: Superiority; p = 1, Regression, Logistic — We used an a priori threshold of p < .05. All 3 comparisons run within same logistic regression model, correcting for the 3 pairwise comparisons using Tukey's Contrasts; Odds Ratio (OR) = 0.9980487, 95% CI 2-sided [0.8680298 to 1.147543]
Statistical Analysis 2: Comparison: Focused on Provider Communication vs Focused on Medical Information Access; Test type: Superiority; p = 0.276, Regression, Logistic — [p-value comment as in outcome 7, analysis 1]; Odds Ratio (OR) = 0.8953032, 95% CI 2-sided [0.7771682 to 1.031395]
Statistical Analysis 3: Comparison: Focused on Scheduling vs Focused on Medical Information Access; Test type: Superiority; p = 0.289, Regression, Logistic — [p-value comment as in outcome 7, analysis 1]; Odds Ratio (OR) = 0.8970536, 95% CI 2-sided [0.7785981 to 1.033531]

8. Secondary Outcome: Link Clicked: Within Less-is-better (Provider Communication vs. Managing Appointments vs. Medical Information Access)
Description: Whether the link / button to start the activation process was clicked (yes / no)
Time Frame: 8-10 days post-intervention
Population: Patients who opened the intervention email and for whom there was a record in the EHR 10 days post-intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Focused on Provider Communication | Focused on Scheduling | Focused on Medical Information Access
Number analyzed (Participants) | 524 | 522 | 482
Participants | 45 | 42 | 73
Statistical Analysis 1: Comparison: Focused on Provider Communication vs Focused on Scheduling; Test type: Superiority; p = 0.94591, Regression, Logistic — [p-value comment as in outcome 7, analysis 1]; Odds Ratio (OR) = 0.9313889, 95% CI 2-sided [0.6003591 to 1.444944]
Statistical Analysis 2: Comparison: Focused on Provider Communication vs Focused on Medical Information Access; Test type: Superiority; p = 0.0041, Regression, Logistic — [p-value comment as in outcome 7, analysis 1]; Odds Ratio (OR) = 1.8998642, 95% CI 2-sided [1.2809137 to 2.817898]
Statistical Analysis 3: Comparison: Focused on Scheduling vs Focused on Medical Information Access; Test type: Superiority; p = 0.0015, Regression, Logistic — [p-value comment as in outcome 7, analysis 1]; Odds Ratio (OR) = 2.0398184, 95% CI 2-sided [1.3648075 to 3.048678]

9. Secondary Outcome: Enrollment: Within Less-is-better (Provider Communication vs. Managing Appointments vs. Medical Information Access)
Description: Whether the patient enrolled in myGeisinger (yes / no)
Time Frame: 8-10 days post-intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Focused on Provider Communication | Focused on Scheduling | Focused on Medical Information Access
Number analyzed (Participants) | 524 | 522 | 482
Participants | 24 | 28 | 31
Statistical Analysis 1: Comparison: Focused on Provider Communication vs Focused on Scheduling; Test type: Superiority; p = 0.829, Regression, Logistic — [p-value comment as in outcome 7, analysis 1]; Odds Ratio (OR) = 1.180837, 95% CI 2-sided [0.6750639 to 2.065546]
Statistical Analysis 2: Comparison: Focused on Provider Communication vs Focused on Medical Information Access; Test type: Superiority; p = 0.404, Regression, Logistic — [p-value comment as in outcome 7, analysis 1]; Odds Ratio (OR) = 1.432003, 95% CI 2-sided [0.8279689 to 2.476702]
Statistical Analysis 3: Comparison: Focused on Scheduling vs Focused on Medical Information Access; Test type: Superiority; p = 0.753, Regression, Logistic — [p-value comment as in outcome 7, analysis 1]; Odds Ratio (OR) = 1.212702, 95% CI 2-sided [0.7161724 to 2.053480]

10. Secondary Outcome: Email Opened: Within Less-is-better (Provider Communication vs. Managing Appointments vs. Medical Information Access)
Description: Whether email was opened (yes / no)
Time Frame: 32-35 days post-intervention
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Focused on Provider Communication | Focused on Scheduling | Focused on Medical Information Access
Number analyzed (Participants) | 2107 | 2094 | 2107
Participants | 568 | 554 | 504
Statistical Analysis 1: Comparison: Focused on Provider Communication vs Focused on Scheduling; Test type: Superiority; p = 0.9284, Regression, Logistic — [p-value comment as in outcome 7, analysis 1]; Odds Ratio (OR) = 0.9747188, 95% CI 2-sided [0.8501783 to 1.1175028]
Statistical Analysis 2: Comparison: Focused on Provider Communication vs Focused on Medical Information Access; Test type: Superiority; p = 0.0612, Regression, Logistic — [p-value comment as in outcome 7, analysis 1]; Odds Ratio (OR) = 0.8518974, 95% CI 2-sided [0.7414610 to 0.9787827]
Statistical Analysis 3: Comparison: Focused on Scheduling vs Focused on Medical Information Access; Test type: Superiority; p = 0.1407, Regression, Logistic — [p-value comment as in outcome 7, analysis 1]; Odds Ratio (OR) = 0.8739930, 95% CI 2-sided [0.7602296 to 1.0047804]

11. Secondary Outcome: Link Clicked: Within Less-is-better (Provider Communication vs. Managing Appointments vs. Medical Information Access)
Description: Whether the link / button to start the activation process was clicked (yes / no)
Time Frame: 32-35 days post-intervention
Population: Patients who opened the intervention email and for whom there was a record in the EHR 32 days post-intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Focused on Provider Communication | Focused on Scheduling | Focused on Medical Information Access
Number analyzed (Participants) | 568 | 554 | 504
Participants | 57 | 51 | 80
Statistical Analysis 1: Comparison: Focused on Provider Communication vs Focused on Scheduling; Test type: Superiority; p = 0.8848, Regression, Logistic — [p-value comment as in outcome 7, analysis 1]; Odds Ratio (OR) = 0.9089673, 95% CI 2-sided [0.6109603 to 1.352333]
Statistical Analysis 2: Comparison: Focused on Provider Communication vs Focused on Medical Information Access; Test type: Superiority; p = 0.0127, Regression, Logistic — [p-value comment as in outcome 7, analysis 1]; Odds Ratio (OR) = 1.6914929, 95% CI 2-sided [1.1762411 to 2.432450]
Statistical Analysis 3: Comparison: Focused on Scheduling vs Focused on Medical Information Access; Test type: Superiority; p = 0.0033, Regression, Logistic — [p-value comment as in outcome 7, analysis 1]; Odds Ratio (OR) = 1.8608951, 95% CI 2-sided [1.2800275 to 2.705356]

12. Secondary Outcome: Enrollment: Within Less-is-better (Provider Communication vs. Managing Appointments vs. Medical Information Access)
Description: Whether the patient enrolled in myGeisinger (yes / no)
Time Frame: 32-35 days post-intervention
Population: Patients who opened the intervention email and for whom there was a record in the EHR 32 days post-intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Focused on Provider Communication | Focused on Scheduling | Focused on Medical Information Access
Number analyzed (Participants) | 568 | 554 | 504
Participants | 54 | 46 | 52
Statistical Analysis 1: Comparison: Focused on Provider Communication vs Focused on Scheduling; Test type: Superiority; p = 0.759, Regression, Logistic — [p-value comment as in outcome 7, analysis 1]; Odds Ratio (OR) = 0.8619131, 95% CI 2-sided [0.5709078 to 1.301251]
Statistical Analysis 2: Comparison: Focused on Provider Communication vs Focused on Medical Information Access; Test type: Superiority; p = 0.897, Regression, Logistic — [p-value comment as in outcome 7, analysis 1]; Odds Ratio (OR) = 1.0950508, 95% CI 2-sided [0.7331329 to 1.635633]
Statistical Analysis 3: Comparison: Focused on Scheduling vs Focused on Medical Information Access; Test type: Superiority; p = 0.498, Regression, Logistic — [p-value comment as in outcome 7, analysis 1]; Odds Ratio (OR) = 1.2704886, 95% CI 2-sided [0.8377249 to 1.926816]

ADVERSE EVENTS:
Time Frame: No adverse events were evaluated.
Description: We only received information about email engagement and portal enrollment. We did not collect or receive any information regarding adverse events.
Arm/Group | Control | Focused on Provider Communication | Focused on Scheduling | Focused on Medical Information Access | Social Proof | Endowment / Decision Staging
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
For this study, we only received data about engagement with the email and enrollment in the patient portal. Demographic information such as age, sex, or gender were not collected. Note that for some patients, enrollment data could not be extracted from Geisinger's electronic health records; these patients were excluded from analyses. Also note that "1 week" and "1 month" outcome data were extracted within a time range that was a few days longer than 7 and 30 days post-intervention, respectively.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-05): https://cdn.clinicaltrials.gov/large-docs/14/NCT04332614/Prot_SAP_000.pdf